### Expanding the Click City Tobacco Prevention Program to Include E-cigarettes and Other Novel Tobacco Products

Request for Passive Consent to Parents and Active Decline Response

NCT 036872900 March 6, 2023

#### Click City Tobacco Project

Dear Parents or Guardians,

Your child's/student's school is participating in a study of a tobacco/e-cigarette prevention program (*Click City Tobacco*) with 5<sup>th</sup> graders. This study is funded by the National Institutes of Health, and is being conducted by the University of Arizona and the Oregon Research Behavioral Intervention Strategies at Oregon Research Institute in Eugene, Oregon.

Students will complete two, 15-minute, on-line surveys (before and after using the *Click City Tobacco* program). The surveys ask questions about the student's attitude toward tobacco use (including cigarettes, e-cigarettes and smokeless tobacco) and tobacco users, their perceptions of risk related to tobacco use, and their intentions to use tobacco in the future. They will also be asked if members of their family use tobacco.

Students will use their state identification numbers on the surveys instead of their name. Researchers will not know the names of the students. All answers will be kept confidential. That means they will not share individual answers with anyone.

Because we want to test how well the *Click City Tobacco* program works, students in half of the participating schools will use the *Click City Tobacco* program while the other half will continue to use their usual tobacco prevention curriculum. After the surveys are completed, all participating schools will receive the program for use for one year.

We are asking for your permission to allow your student to participate in answering our surveys. If you do not want your student to participate, complete and return the enclosed form in the stamped envelope by mail. If we do not hear from you, we will assume that you agree to have your child/student complete our surveys.

Completing our surveys is voluntary, and parents can choose not to have their 5<sup>th</sup> grader participate at any time during the study. Your child's/student's grade or their relationship with their teacher will not be affected if they do not participate in the study.

If you have any questions or concerns, please call Jessica Olson at (541) 484-2123, ext. 2149 or Yessenya Barraza at (520) 626-9291. We hope you will join us in making this project a success.

Sincerely,

#### El Proyecto de Click City sobre Tabaco

Queridos padres,

Estamos estudiando un programa de prevención de tabaco/cigarrillos electrónicos (Click City Tabaco) con alumnos de 5to grado en la escuela de su hijo(a)/estudiante. Este estudio está financiado por el Instituto Nacional de Salud y esta llevado a cabo por Innovaciones Influyentes en el Instituto de Oregón de Investigaciones en Eugene, Oregón y la Universidad de Arizona en Tucson, Arizona.

Los estudiantes completaran dos encuestas en línea de 15 minutos (antes y después de completar el programa Click City Tabaco). Las encuestas hacen preguntas sobre la actitud del estudiante hacia el consumo de tabaco (incluyendo los cigarrillos, los cigarrillos electrónicos y el tabaco sin humo) y sobre los consumidores de tabaco, sus percepciones del riesgo relacionado con el consumo de tabaco y sus intenciones de consumirlo en el futuro. También se les preguntara si los miembros de su familia usan el tabaco.

Los estudiantes usaran sus números de identificación estatales en las encuestas en lugar de su nombre. No se identificara los nombres de los estudiantes. Todas las respuestas se mantendrán confidenciales. Eso significa que no compartiremos respuestas individuales con nadie.

Debido a que queremos evaluar que tan bien funciona el programa *Click City Tabaco*, la mitad de los estudiantes de las escuelas participantes usaran el programa *Click City Tabaco* mientras la otra mitad continuara usando su currículum de estudios habitual de prevención del tabaco.

Le pedimos su permiso para permitir que su estudiante participe en nuestras encuestas. Si no desea que su estudiante participe, por favor complete y devuelva el formulario adjunto en el sobre sellado por correo. Si no tenemos noticias suyas, asumiremos que acepta que su hijo(a)/estudiante complete nuestras encuestas.

Es voluntario completar nuestras encuestas, y los padres pueden optar su hijo(a) de 5to grado que no participe en ningún momento durante el estudio. La calificación de su hijo(a)/estudiante o su relación con su maestro(a) no serán afectadas si no participan en el estudio.

Si tiene alguna pregunta o duda llame a Jessica Olson en Innovaciones Influyentes al (541) 484-2123, ext. 2149, o Yessenya Barraza en la Universidad de Arizona al (520) 626-9291. Esperemos que se una a nosotros para que este proyecto sea un éxito.

Sinceramente.

### [INSERT SCHOOL NAME HERE]

## Passive Consent form for parents of students in the effectiveness study

IF YOU DO NOT WANT YOUR STUDENT TO PARTICIPATE, COMPLETE AND RETURN THE ENCLOSED FORM IN THE STAMPED ENVELOPE BY MAIL BY [DATE].

I understand that completing and returning this form indicates that I **do not** want my 5<sup>th</sup> grader to complete the *Click City Tobacco* program surveys.

| I do not want my child to complete the Click City Tobacco program (Please check box) | m surveys. |
|---|---|
| Child's Name (First and Last) | |
| Child's Birthday (Month and Day only) | |
| Child's School | |
| Parent or Guardian Signature | |
| Date | |

PUT STUDENT ID LABEL HERE

### [INSERT SCHOOL NAME HERE]

# Formulario de consentimiento pasivo para padres de jóvenes en el estudio de efectividad

SI NO DESEA QUE SU ESTUDIANTE PARTICIPE, POR FAVOR COMPLETE Y DEVUELVA EL FORMULARIO ADJUNTO EN EL SOBRE SELLADO POR CORREO ANTES DEL [FECHA].

Entiendo que completar y devolver este formulario indica que **no le doy permiso** a mi hijo(a) de 5to grado que complete las encuestas del programa *Click City Tabaco*.

| Tiljo(a) de 5to grado que complete las chodestas del programa eller el | ty rabacc. |
|---|---|
| No le doy permiso a mi hijo(a) que complete las encuestas del p<br>City Tabaco. (Marque la casilla) | rograma Click |
| Nombre del joven (nombre y apellido) | |
| Fecha de Nacimiento del joven (mes y día solamente) | |
| Escuela del joven | |
| Firma del padre o tutor | |
| Fecha | |

PUT STUDENT ID LABEL HERE